CLINICAL TRIAL: NCT00444444
Title: Clinical Analysis for Predicting of Relapse During Steroid Treatment for Autoimmune Pancreatitis (AIP) in Korean Population Based on the HLA Analysis by Using a High Resolution (Sequence Based) Techniques
Brief Title: Genetic Analysis for Predicting of Relapse During Steroid Treatment for Autoimmune Pancreatitis (AIP)
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Other Study IDs: 2007-0038
Record Dates: First submitted 2007-03-06; First posted 2007-03-07 (Estimated); Last update posted 2007-06-26 (Estimated); Status verified 2007-03

CONDITIONS: Pancreatitis
Keywords: Autoimmune pancreatitis, HLA, relapse, Sequence-based typing
MeSH Terms: conditions — Pancreatitis; Autoimmune Pancreatitis; Recurrence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To determine whether certain alleles or haplotypes of major histocompatibility complex gene are associated with AIP in Korean population, we undertook this study with high-resolution typing for HLA (sequence-based typing).

Primary outcomes: detection of novel allele associated with AIP in Korean population Secondary outcomes: detection of genetic factor for relapse of AIP during steroid treatment

DETAILED DESCRIPTION:
Autoimmune chronic pancreatitis (AIP) can be defined as a chronic inflammation of the pancreas due to an autoimmune mechanism; autoimmunity is responsible for producing the pancreatic lesion. AIP is a distinctive type of chronic pancreatitis that shows reversible improvement of pancreatic morphology and function with oral steroid therapy, in comparison to other types of chronic pancreatitis which hardly respond to various treatments. AIP is increasingly being recognized to be a worldwide entity. The sudden increment in cases reported probably reflects the growing awareness of the entity, rather than a rise in the true incidence. In previous Japanese report, HLA DRB1*0405-DQB*0401 haplotype may be associated with autoimmune pancreatitis in the Japanese population. However, to date there was no subsequent data for supporting these results. In addition, this Japanese study had a limitation in methodology by using a low-resolution typing for HLA. Although this entity is well responsive to steroid therapy, relapse of AIP during steroid treatment is not uncommon. Unfortunately, there has been no laboratory or genetic predictor for responsiveness to steroid therapy in patients with AIP. To further clarify and confirm high-risk and protective genotypes for autoimmune diseases, therefore, high-resolution typing for HLA should be needed. Thus, to determine whether certain alleles or haplotypes of major histocompatibility complex gene are associated with AIP in Korean population, we undertook this study with high-resolution typing for HLA (sequence-based typing).

ELIGIBILITY:
Inclusion Criteria:

* Patient with autoimmune pancreatitis
* The diagnosis is mainly based on the following three characteristic findings proposed by Japan Pancreas Society in 2002: (1)Imaging studies: irregular narrowing of the main pancreatic duct and diffuse enlargement of the pancreas, (2) Laboratory data: elevated serum IgG or the presence of autoantibodies, (3) Histological examinations: fibrotic changes with lymphoplasmacytic infiltration in the pancreatic tissue.
* Age 18 years and above
* No serious medical or psychological condition that would preclude study treatment
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures

Exclusion Criteria:

* Age below 18 years
* Pregnancy
* Active alcohol or drug abuse
* Unstable or unwilling to comply with follow up

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2002-02; Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Do Hyun Park, MD, PhD, Study Director — Soon Chun Hyang University; Myung-Hwan Kim, MD, PhD, Study Chair — Asan Medical Center
Locations (1):
- Department of Internal Medicine, University of Ulsan College of Medicine, Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Park DH, Kim MH, Oh HB, Kwon OJ, Choi YJ, Lee SS, Lee TY, Seo DW, Lee SK. Substitution of aspartic acid at position 57 of the DQbeta1 affects relapse of autoimmune pancreatitis. Gastroenterology. 2008 Feb;134(2):440-6. doi: 10.1053/j.gastro.2007.11.023. Epub 2007 Nov 17. PMID 18155707